CLINICAL TRIAL: NCT05872906
Title: Using Ultrasound and Acupuncture to Explore the De-qi Location and Reaction of Specific Acupoints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CMUH112-REC2-016
Record Dates: First submitted 2023-04-21; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: de qi of Acupuncture; Ultrasound Imaging
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupuncture (Experimental): All subjects will receive acupuncture at LI11, ST36, SP10, SP9, SP6, ST34, BL39, KI10, LIV8, LI10, HT3, SI8, LI4, PC6, HT7, GB34, GB40, KI3, BL2, GB20, LIV3, BL62, KI6, BI57, ST40, KI7 and be recorded with simultaneous ultrasound imaging, external video, and required to fill out sensation sheets. Pulse diagnosis will be taken after de qi is achieved.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — A 1.5-inch needle of 34 gauge (CASOON stainless steel acupuncture needles) is inserted. The physician will then locate the de qi location of the test subjects and elicit a de qi response accompanied by muscle twitch.

SUMMARY:
According to ancient literature, when de qi occurs in the process of acupuncture, the patient may experience sensations such as soreness, numbness, heaviness, swelling. Meanwhile, the acupuncturist may experience the sensation of "a fish taking a bite from the bait on a hook". However, for a beginner at acupuncture, before they have learned to trigger the de qi sensation, it is hard for them to learn according to the ambiguous definition of "a fish taking a bite from the bait on a hook" and thus hard to know whether they have reached the correct location and stimulated de-qi. In this study, through multiple experienced acupuncturists acupuncture multiple test subjects, the investigators will locate the location and the reaction of de qi on the acupoint Quchi (LI11) with ultrasound observation and recording. Through the ultrasound teaching and guidance, the investigators will test whether it is possible to reversely use ultrasound imaging to guide less experienced acupuncturists to the de qi location and elicit de qi response on multiple test subjects. Therefore, the investigators propose this study to test the following hypothesis:"There is a specific anatomical site where de qi occurs at LI11, and it is possible to use ultrasound imaging to guide learners to reach that location and trigger de-qi and that it is applicable to other acupoints". To explore the above hypothesis, the investigators will target the following specific aims. Aim 1: Use ultrasound record and indicate the precise anatomical location and reaction when de qi occurs on acupoint LI11. Aim 2: Simultaneously record the physicians' needling sensations, the participants' needling sensations, twitch response of the participant under ultrasound images. Aim 3: Prove the feasibility of using ultrasound to guide inexperienced physicians to reach the correct location and elicit de qi sensation on the participants. Aim 4: Discuss the relationship between de qi and pulse diagnosis. Aim 5: Apply the above procedures to other acupuncture points such as LU5(Chize), PC3 (Quze),…etc.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20 years and healthy subjects

Exclusion Criteria:

* pregnancy
* patients with chronic diseases such as hypertension, diabetes mellitus, chronic hepatitis, chronic kidney disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-03-05 (Estimated); Study Completion 2024-03-05 (Estimated)

PRIMARY OUTCOMES:
B-mode ultrasound image of the acupuncture site using a linear probe | during each needling process of all acupuncture points over a course of 12 weeks
  B-mode ultrasound image of the acupuncture site using a linear probe will be recorded throughout the needling process. The video would enable the investigators to identify the underlying anatomical structures of the acupuncture point and locate the location of the needle tip where de qi occurs.
Subject sensation questionnaire modified from the Massachusetts General Hospital Acupuncture Sensation Scale (MASS) | during each needling process of all acupuncture points over a course of 12 weeks
  Needling sensations will be collected throughout the needling process.
Subject sensation questionnaire modified from the Southampton Needle Sensation Questionnaire (SNSQ) | during each needling process of all acupuncture points over a course of 12 weeks
  Needling sensations will be collected throughout the needling process.
Pulse wave data taken with ANSWatch | immediately prior to (within 5 minutes) and after (within 5 minutes) needling of each acupuncture point over a course of 12 weeks
  Pulse wave data will be taken with ANSWatch. Data for each test subject will be collected prior to and after the needling process (de qi is achieved).
External video footage of visually observable events (such as muscle contraction) associated with de qi event | during each needling process of all acupuncture points over a course of 12 weeks
  An external video footage will be recorded of the acupuncture site during the needling process

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No